CLINICAL TRIAL: NCT02728466
Title: Investigation on the Effects of Cocoa Procyanidins on Vascular Function in Healthy Individuals
Brief Title: Effects of Cocoa Procyanidins on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Cocoa procyanidins; 12-018 (Other: CTSU)
Record Dates: First submitted 2016-03-09; First posted 2016-04-05 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: flavanols; cocoa procyanidins; vascular function; endothelial function
MeSH Terms: interventions — Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flavanol and procyanidin supplement (Active Comparator): Sustained intake (2x daily over 1 month) of a cocoa-based supplement containing flavanols (monomers) and procyanidins (dimers to decamers)
  Interventions: Dietary Supplement: Flavanol and procyanidin supplement
- Procyanidin-containing supplement (Active Comparator): Sustained intake (2x daily over 1 month) of a cocoa-based supplement containing procyanidins (dimers to decamers)
  Interventions: Dietary Supplement: Procyanidin-containing supplement
- Flavanols and procyanidins deprived supplement (Placebo Comparator): Control supplement deprived of flavanols and procyanidins Sustained intake (2x daily over 1 month) of a macro-and micronutrient matched supplement
  Interventions: Dietary Supplement: control supplement deprived of flavanols and procyanidins

INTERVENTIONS:
Dietary Supplement: Flavanol and procyanidin supplement — Sustained intake (2x daily over 1 month) of a cocoa-based supplement containing flavanols (monomers) and procyanidins (dimers to decamers)
  Arms: Flavanol and procyanidin supplement
Dietary Supplement: Procyanidin-containing supplement — Sustained intake (2x daily over 1 month) of a cocoa-based supplement containing procyanidins (dimers to decamers)
  Arms: Procyanidin-containing supplement
Dietary Supplement: control supplement deprived of flavanols and procyanidins — Placebo comparator: flavanol and procyanidin deprived supplement Sustained intake (2x daily over 1 month) of a macro-and micronutrient matched supplement
  Arms: Flavanols and procyanidins deprived supplement

SUMMARY:
There is a question regarding the role of higher flavanol oligomers (procyanidins) and of intestinal flavanol metabolites i.e. valerolactones, in the context of flavanol intake-related vascular effects. Only flavanol monomers, and to a certain degree dimers, are absorbed in the small intestine and enter circulation. Higher oligomers (procyanidins) are not absorbed and are catabolized by the colonic microflora. The catabolites enter the circulation. Phenolic acids and valerolactones represent a significant proportion of these catabolites, reaching peak concentrations in the order of 6-10 h post ingestion. The vascular effects of these colonic microbiome-derived flavanol derivatives have not been studied so far. The purpose of the study is to determine the timecourse of endothelial function along with flavanol catabolites & metabolites during acute, sustained, and acute on sustained ingestion of procyanidins as compared to previously used flavanol interventions, and flavanol free control.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects (no clinical signs or symptoms of cardiovascular disease)
* >18 years, <35 years

Exclusion Criteria:

* cardiovascular disease
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* C-reactive protein > 1 mg/dl
* malignant disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change form Baseline Endothelial function at 1 month | Baseline and 1 month
  Measured by Flow mediated dilation (FMD) at 0 and 2 hours postconsumption on baseline and on 1 month

SECONDARY OUTCOMES:
Plasma flavanol metabolites | Baseline and 1 month
  Measured by high performance liquid chromotography (HPLC) at 2 hours and on 1 month postconsumption
Urinary flavanol metabolites | Baseline and 1 month
  Measured up to 24 hours post consumption on day 1 and 1 month after consumption
Urinary valerolactone metabolites | Baseline and 1 month
  Measured up to 24 hours post consumption on day 1 and 1 month after consumption

OTHER OUTCOMES:
Pulse wave velocity | Baseline and 1 month
  Measured by SphygmoCor on baseline 2 hours postconsumption and on 1 month.
Blood pressure | Baseline and 1 month
  automatical measurements on baseline 2 hours postconsumption and on 1 month
high density lipoproteins (HDL) | Baseline and 1 month
  measured on baseline and after 1 month
low density lipoproteins (LDL) | Baseline and 1 month
  measured on baseline and after 1 month
cholesterol | Baseline and 1 month
  measured on baseline and after 1 month
triglyceride | Baseline and 1 month
  measured on baseline and after 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiß, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf; Malte Kelm, Prof. MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Mateos A, Weber T, Skene SS, Ottaviani JI, Crozier A, Kelm M, Schroeter H, Heiss C. Assessing the respective contributions of dietary flavanol monomers and procyanidins in mediating cardiovascular effects in humans: randomized, controlled, double-masked intervention trial. Am J Clin Nutr. 2018 Dec 1;108(6):1229-1237. doi: 10.1093/ajcn/nqy229. PMID 30358831